CLINICAL TRIAL: NCT06806410
Title: The Efficacy of Liposomal Bupivacaine in Ultrasound Guided Supraclavicular Nerve Blocks for Hand and Wrist Surgery: a Prospective, Randomized, Blinded Controlled Trial
Brief Title: The Efficacy of Liposomal Bupivacaine in Ultrasound Guided Supraclavicular Nerve Blocks for Hand and Wrist Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLIR2023-34
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Hand Surgery; Wrist Surgery; Elbow Surgery; Fracture Fixation; Dupuytren Contracture; Finger Fracture; Wrist Arthropathy; Distal Radius Fracture
Keywords: liposomal bupivacaine; supraclavicular nerve block; ultrasound guided nerve block; hand, wrist, elbow surgery; local anesthetic; dexamethasone perineural injection
MeSH Terms: conditions — Dupuytren Contracture; Wrist Fractures | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: randomization into three groups. Control group is administration of local anesthesia in ultrasound guided supraclavicular nerve blocks. There are two study groups. The intermediate study group is administration of local anesthesia with dexamethasone in the ultrasound guided supraclavicular nerve block. The other study group is administration of liposomal bupivacaine in the ultrasound guided supraclavicular nerve block.
Who Masked: Participant
Masking Description: the patient is blinded to the study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Arm: local anesthesia only in ultrasound guided supraclavicular nerve block (No Intervention): ultrasound guided supraclavicular nerve blocks are typically performed with the use of local anesthesia only
- Study Arm: local anesthesia with perineural dexamethasone (Experimental): dexamethasone is a potent steroid that when provided in ultrasound guided nerve blocks can extend the duration of the nerve block.
  Interventions: Drug: Dexamethasone
- Study Arm: liposomal bupivacaine (Experimental): our study team would like to determine how use of liposomal bupivacaine in supraclavicular nerve blocks can lengthen the duration of the nerve block, and how it may affect the number of opioid pills used after surgery up until postoperative day three.
  Interventions: Drug: Liposomal bupivacaine (LB)

INTERVENTIONS:
Drug: Liposomal bupivacaine (LB) — our study team wishes to determine effect of liposomal bupivacaine in regional nerve blocks for surgery of the upper extremity (finger, hand, wrist, elbow)
  Other Names: liposomal bupivacaine; exparel
  Arms: Study Arm: liposomal bupivacaine
Drug: Dexamethasone — dexamethasone injected in perineural area can extend the regional nerve block
  Other Names: decadron perineural injection
  Arms: Study Arm: local anesthesia with perineural dexamethasone

SUMMARY:
Patients undergoing hand, wrist, and elbow surgery may experience pain after surgery. The orthopedic surgeon may provide prescription pain medications after surgery to assist with pain control. However, with concern of the opioid epidemic, many patients would rather minimize the use of narcotic pain prescriptions after having surgery. As an alternative, ultrasound guided regional nerve blocks can assist with postoperative pain control.

patients consented to this study will be randomized into three groups: 1) will receive an ultrasound guided nerve block with local anesthesia only, 2) will receive an ultrasound guided nerve block with local anesthesia and a steroid dexamethasone, 3) will receive an ultrasound guided nerve block with liposomal bupivacaine.

our study team will make phone calls after surgery to the patient to determine how long the block lasted for, and how many opioid pain pills were taken up to 3 days after surgery.

DETAILED DESCRIPTION:
Our study team predicts that the ultrasound guided nerve block with liposomal bupivacaine can last approximately 48 hours, while the block with local anesthesia and dexamethasone will last approximately 30 hours, and the block with local anesthesia only may last up to 24 hours

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo finger, hand, wrist, elbow surgery with a hand surgeon at St. Luke's University Hospital in Bethlehem, Pennsylvania
* patients greater than 18 years of age, able to provide written consent for surgery and study

Exclusion Criteria:

* patients that cannot provide written consent for finger, hand, wrist, elbow surgery
* patients with known allergies to local anesthetics
* patients with severe liver disease
* patients with a condition known as methemoglobinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Subjective length of duration of block | feedback obtained up until day 3 after surgery
  our study team contacts the patients 4 days after surgery to ask how long their regional nerve block lasted

SECONDARY OUTCOMES:
Number of opioid pills taken until postoperative day 3 | feedback until day 3 after surgery
  our study team contacts the patients to ask how many opioid pain pills were taken from arrival to home up until postoperative day 3

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ng-Pellegrino, MD, Principal Investigator — St. Luke's Hospital and Health Network, Pennsylvania
Locations (1):
- St. Luke's University Health Network, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
we will provide results on our measured outcomes: subjective length of duration of block, number of opioid pills taken by postsurgical day 3. we will provide de-identified information on demographics as well between the control arm and treatment arms
Supporting Information: Study Protocol, SAP, CSR
Time Frame: we will provide deidentified data on patients participating within the start to end dates of patient recruitment. This data will be available to view in anticipated publication to a journal
Access Criteria: This information can be available to view after publication to a journal.